CLINICAL TRIAL: NCT02401230
Title: Defining the Rectal Mucosa in Men Who Have Sex With Men at Risk of HIV Infection
Brief Title: PrEP, Lube, and the Rectal Mucosa in MSM at Risk of HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00077593
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-12

CONDITIONS: HIV
Keywords: Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome Virus; Pre-exposure Prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Rectal Gel Lubricant (Active Comparator): Subjects will insert 5 mL of lubricant in rectum for seven consecutive days
  Interventions: Device: Gel lubricant
- Truvada (Active Comparator): Subjects will take one Truvada tablet orally for seven consecutive days
  Interventions: Drug: Truvada
- Rectal Gel Lubricant + Truvada (Active Comparator): Subjects will insert 5 mL of lubricant in rectum and take one Truvada tablet orally for seven consecutive days
  Interventions: Drug: Truvada; Device: Gel lubricant

INTERVENTIONS:
Drug: Truvada — Truvada is a combination of 200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate taken orally.
  Other Names: Emtricitabine; Tenofovir
  Arms: Rectal Gel Lubricant + Truvada; Truvada
Device: Gel lubricant — Five ml of an over the counter sexual lubricant will be dispensed using an applicator.
  Arms: Rectal Gel Lubricant; Rectal Gel Lubricant + Truvada

SUMMARY:
The purpose of this study is to determine whether the use of rectal lubricants can affect how well the medication, Truvada, will work to prevent infection with HIV when someone is exposed to HIV in the rectum.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) continue to be disproportionately affected by HIV. The majority of HIV infections among MSM occur through exposure to the rectal mucosa during receptive anal intercourse (RAI). During RAI, many MSM will use lubricants, which can potentially cause mucosal inflammation and damage. A new HIV prevention intervention, called pre-exposure prophylaxis (PrEP), recommends that MSM at risk of HIV infection take a daily anti-HIV medication called Truvada (tenofovir/emtricitabine) which is highly effective. However, it is not known if the use of lubricant during RAI will interfere with the efficacy of PrEP for HIV prevention.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative man who reports receptive anal sex with another man in the last 6 months aged 18-49 years
* Male to female transgender women who are not currently taking hormonal therapy or plan to take hormonal therapy for the duration of the study
* Not currently taking pre-exposure prophylaxis (PrEP) and no plans to initiate during study
* Able to provide informed consent in English
* No plans for relocation in the next 6 months
* Willing to undergo peripheral blood and rectal biopsy sampling
* Willing to use study products as directed
* Willing to abstain from receptive anal intercourse 3 days prior to study visit 2 (4-16 weeks after the screening visit)and 10 days prior to study visit 4 (5-26 weeks after the screening visit)
* Willing to abstain from receptive anal intercourse for 1 week after study visit 2 (4-16 weeks after the screening visit) and study visit 4 (5-26 weeks after the screening visit)

Exclusion Criteria:

* History of inflammatory bowel disease or other inflammatory, infiltrative, infectious or vascular condition involving the lower gastrointestinal tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel
* Significant laboratory abnormalities at baseline visit for rectal biopsies, including but not limited to:

  1. Hemoglobin (Hbg) ≤ 10 g/dL
  2. Partial thromboplastin time (PTT) > 1.5x upper limit normal (ULN) or international normalized ratio (INR) > 1.5x ULN
  3. Platelet count <100,000
* Any known medical condition that, in the judgment of the investigators, increases the risk of local or systemic complications of endoscopic procedures or pelvic examination, including but not limited to:

  1. Uncontrolled or severe cardiac arrhythmia
  2. Recent major abdominal, cardiothoracic, or neurological surgery
  3. History of uncontrolled bleeding diathesis
  4. History of colonic, rectal, or vaginal perforation, fistula, or malignancy
  5. History or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the anorectal or vaginal mucosa, or untreated sexually transmitted disease with mucosal involvement
* Continued need for, or use during the 14 days prior to enrollment, of the following medications:

  1. Aspirin or more than 4 doses of nonsteroidal anti-inflammatory drugs (NSAIDs)
  2. Warfarin, heparin (low-molecular weight or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
  3. Any form of rectally administered agent besides products lubricants or douching used for sexual intercourse
* Continued need for, or use during the 90 days prior to enrollment, of the following medications:

  1. Systemic immunomodulatory agents
  2. Supraphysiologic doses of steroids
  3. Experimental medications, vaccines, or biologicals
* Intent to use HIV antiretroviral PrEP during the study, outside of the study procedures
* Symptoms of an untreated rectal sexually transmitted infection (e.g. rectal pain, discharge, bleeding, etc.)
* Current use of hormonal therapy
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD/MPH, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of of Emory University, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited March 2015 through November 2016.
Pre-assignment Details: Of the 86 subjects consented for study participation, 76 were randomized to a study intervention.
Groups:
- Rectal Gel Lubricant: Subjects inserted 5 mL of lubricant in rectum for seven consecutive days.
  Gel lubricant: Five ml of an over the counter sexual lubricant will be dispensed using an applicator.
- Truvada: Subjects took one Truvada tablet orally for seven consecutive days.
  Truvada: Truvada is a combination of 200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate taken orally.
- Rectal Gel Lubricant + Truvada: Subjects inserted 5 mL of lubricant in rectum and took one Truvada tablet orally for seven consecutive days
  Truvada: Truvada is a combination of 200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate taken orally.
  Gel lubricant: Five ml of an over the counter sexual lubricant will be dispensed using an applicator.
Period: Overall Study
Arm/Group | Rectal Gel Lubricant | Truvada | Rectal Gel Lubricant + Truvada
Started | 26 | 25 | 25
Completed | 20 | 19 | 21
Not Completed | 6 | 6 | 4
Not completed — Adverse Event | 3 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Participants who began a study intervention and completed all study visits.
Groups:
- Rectal Gel Lubricant: Subjects inserted 5 mL of lubricant in rectum for seven consecutive days
  Gel lubricant: Five ml of an over the counter sexual lubricant will be dispensed using an applicator.
- Truvada: Subjects took one Truvada tablet orally for seven consecutive days
  Truvada: Truvada is a combination of 200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate taken orally.
- Total: Total of all reporting groups
Arm/Group | Rectal Gel Lubricant | Truvada | Rectal Gel Lubricant + Truvada | Total
Number analyzed (Participants) | 20 | 19 | 21 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 21 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 19 | 21 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 21 | 60

OUTCOME MEASURES:

1. Primary Outcome: Median Percentage of CD4 Positive T-Cells
Description: HIV target cell availability will be assessed by the median percentage of CD4+ T cells that express HIV co-receptor CCR5 as measured prior to product use and on day 8 after product use.
Time Frame: Baseline, Post-Intervention (Day 8)
Population: The analysis population includes participants for whom the assay could be accurately performed. Data were not available for analysis in the case of an insufficient sample to perform this assay, poor performance of the assay, or technical issues in the laboratory.
Measure: Median (Inter-Quartile Range); unit: percentage positive T-cells
Arm/Group | Rectal Gel Lubricant | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 10 | 6 | 10
percentage positive T-cells
  Baseline | 62 [50 to 70] | 70 [39 to 76] | 58 [32 to 67]
  Day 8 | 66 [29 to 72] | 58 [39 to 71] | 51 [14 to 61]

2. Primary Outcome: Median Cumulative Amount of p24
Description: The median cumulative amount of p24 produced in a rectal explant challenge assay as measured by ELISA from participants prior to product use and on day 8 after product use.
Time Frame: Baseline, Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Rectal Gel Lubricant | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 4 | 8 | 5
pg/mL
  Baseline | 250 [138 to 608] | 287 [80 to 944] | 276 [82 to 786]
  Day 8 | 363 [102 to 494] | 133 [68 to 363] | 284 [114 to 369]

3. Secondary Outcome: Median Plasma Emtricitabine (FTC) Concentration
Description: Median plasma FTC concentration as measured in ng/ml prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
ng/ml | 248 [71 to 277] | 340 [8 to 509]

4. Secondary Outcome: Median Plasma Tenofovir (TDF) Concentration
Description: Median plasma TDF concentration as measured in ng/ml prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
ng/ml | 52 [27 to 73] | 64 [17 to 87]

5. Secondary Outcome: Median Rectal Secretion Emtricitabine (FTC) Concentration
Description: Median rectal secretions FTC concentrations as measured in ng/swab prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: ng/swab
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
ng/swab | 320 [43 to 661] | 382 [38 to 570]

6. Secondary Outcome: Median Rectal Secretion Tenofovir (TDF) Concentration
Description: Median rectal secretions TDF concentrations as measured in ng/swab prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: ng/swab
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
ng/swab | 812 [170 to 1535] | 780 [61 to 3160]

7. Secondary Outcome: Median Peripheral Blood Mononuclear Cell (PBMC) Emtricitabine (FTC) Concentration
Description: Median blood PBMC FTC concentrations as measured in fmol/million cells prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/million cells
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/million cells | 4980 [1554 to 5730] | 4020 [1399 to 5370]

8. Secondary Outcome: Median Peripheral Blood Mononuclear Cell (PBMC) Tenofovir (TDF) Concentration
Description: Median blood PBMC TDF concentrations as measured in fmol/million cells prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/million cells
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/million cells | 45 [25 to 57] | 48 [24 to 62]

9. Secondary Outcome: Median Rectal Tissue Emtricitabine (FTC) Concentration
Description: Median rectal tissue FTC concentrations as measured in fmol/mg tissue prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/mg tissue
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/mg tissue | 104 [4 to 203] | 112 [16 to 137]

10. Secondary Outcome: Median Rectal Tissue Tenofovir (TDF) Concentration
Description: Median rectal tissue TDF concentrations as measured in fmol/mg tissue prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/mg tissue
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/mg tissue | 510 [4 to 1191] | 280 [19 to 561]

11. Secondary Outcome: Median Rectal Tissue Deoxyadenosine Triphosphate (dATP) Concentration
Description: Median rectal tissue dATP concentrations as measured in fmol/mg tissue prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Baseline, Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/mg tissue
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/mg tissue
  Baseline | 131 [12 to 262] | 74 [19 to 200]
  Post-Intervention (Day 8) | 60 [14 to 155] | 66 [19 to 134]

12. Secondary Outcome: Median Rectal Tissue Deoxycytidine Triphosphate (dCTP) Concentration
Description: Median rectal tissue dCTP concentrations as measured in fmol/mg tissue prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Baseline, Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/mg tissue
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/mg tissue
  Baseline | 246 [7 to 414] | 58 [10 to 395]
  Post-Intervention (Day 8) | 43 [6 to 131] | 36 [11 to 97]

13. Secondary Outcome: Median Peripheral Blood Mononuclear Cell (PBMC) Deoxyadenosine Triphosphate (dATP) Concentration
Description: Median blood dATP concentrations as measured in fmol/million cells prior to product use and on day 8 after product use. The higher the concentration, the better the drug distribution.
Time Frame: Baseline, Post-Intervention (Day 8)
Population: Number of participants who provided a viable sample.
Measure: Median (Inter-Quartile Range); unit: fmol/million cells
Arm/Group | Truvada | Rectal Gel Lubricant + Truvada
Number analyzed (Participants) | 19 | 21
fmol/million cells
  Baseline | 149 [16 to 187] | 140 [25 to 221]
  Post-Intervention (Day 8) | 204 [56 to 269] | 122 [35 to 238]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout study duration (1 year and 7 months).
Arm/Group | Rectal Gel Lubricant | Truvada | Rectal Gel Lubricant + Truvada
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 4/20 | 2/19 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rectal Gel Lubricant (N=20) | Truvada (N=19) | Rectal Gel Lubricant + Truvada (N=21)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT02401230/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT02401230/SAP_001.pdf